CLINICAL TRIAL: NCT07176182
Title: An Open-Label, Two-Arm, Phase II Clinical Trial of Neoadjuvant mFOLFOX (Leucovorin, Fluorouracil, Oxaliplatin) Combined With Citrus Flavonoid Tablets (Alvenor) for Locally Advanced Rectal Cancer Patients With High YWHAB Expression
Brief Title: Clinical Trial of Neoadjuvant mFOLFOX Plus Alvenor for LARC Patients With High YWHAB Expression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2025123
Record Dates: First submitted 2025-08-27; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-05

CONDITIONS: Rectal Cancer Patients; Rectal Cancer Stage II; Rectal Cancer Stage III
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: The trial evaluates a regimen combining mFOLFOX chemotherapy with citrus flavonoid tablets (Alvenor) for neoadjuvant therapy (pre-surgery) and postoperative adjuvant therapy.
  Treatment Protocol
  Preoperative (4-6 cycles) and Postoperative (6-8 cycles):
  Each 14-day cycle includes:
  Oxaliplatin: 85 mg/m² via 180-minute intravenous infusion on Day 1.
  Leucovorin: 400 mg/m² via 120-minute intravenous infusion on Day 1.
  5-Fluorouracil: 2400 mg/m² via continuous intravenous infusion over 46 hours.
  Citrus flavonoid tablets (Alvenor): 500 mg orally three times daily (Days 1-14), administered with or without the chemotherapy regimen (depending on group assignment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mFOLFOX regimen neoadjuvant therapy group (Active Comparator): The trial evaluates a regimen combining mFOLFOX chemotherapy with citrus flavonoid tablets (Alvenor) for neoadjuvant therapy (pre-surgery) and postoperative adjuvant therapy.
  Treatment Protocol
  Preoperative (4-6 cycles) and Postoperative (6-8 cycles):
  Each 14-day cycle includes:
  Oxaliplatin: 85 mg/m² via 180-minute intravenous infusion on Day 1.
  Leucovorin: 400 mg/m² via 120-minute intravenous infusion on Day 1.
  5-Fluorouracil: 2400 mg/m² via continuous intravenous infusion over 46 hours.
  Interventions: Drug: mFOLFOX regimen neoadjuvant therapy group
- mFOLFOX regimen combined with Citrus Flavone Tablets (Alvenor) neoadjuvant treatment group (Experimental): The trial evaluates a regimen combining mFOLFOX chemotherapy with citrus flavonoid tablets (Alvenor) for neoadjuvant therapy (pre-surgery) and postoperative adjuvant therapy.
  Treatment Protocol
  Preoperative (4-6 cycles) and Postoperative (6-8 cycles):
  Each 14-day cycle includes:
  Oxaliplatin: 85 mg/m² via 180-minute intravenous infusion on Day 1.
  Leucovorin: 400 mg/m² via 120-minute intravenous infusion on Day 1.
  5-Fluorouracil: 2400 mg/m² via continuous intravenous infusion over 46 hours.
  Citrus flavonoid tablets (Alvenor) : 500 mg orally three times daily (Days 1-14), administered with or without the chemotherapy regimen (depending on group assignment).
  Interventions: Drug: mFOLFOX regimen combined with Citrus Flavone Tablets (Alvenor) neoadjuvant treatment group

INTERVENTIONS:
Drug: mFOLFOX regimen combined with Citrus Flavone Tablets (Alvenor) neoadjuvant treatment group — The trial evaluates a regimen combining mFOLFOX chemotherapy with citrus flavonoid tablets (Alvenor) for neoadjuvant therapy (pre-surgery) and postoperative adjuvant therapy.
  Treatment Protocol
  Preoperative (4-6 cycles) and Postoperative (6-8 cycles):
  Each 14-day cycle includes:
  Oxaliplatin: 85 mg/m² via 180-minute intravenous infusion on Day 1.
  Leucovorin: 400 mg/m² via 120-minute intravenous infusion on Day 1.
  5-Fluorouracil: 2400 mg/m² via continuous intravenous infusion over 46 hours.
  Citrus flavonoid tablets (Alvenor) : 500 mg orally three times daily (Days 1-14), administered with or without the chemotherapy regimen (depending on group assignment).
  Other Names: 5-Fluorouracil, Oxaliplatin, Citrus Flavone Tablets (Alvenor)
  Arms: mFOLFOX regimen combined with Citrus Flavone Tablets (Alvenor) neoadjuvant treatment group
Drug: mFOLFOX regimen neoadjuvant therapy group — The trial evaluates a regimen combining mFOLFOX chemotherapy with citrus flavonoid tablets (Alvenor) for neoadjuvant therapy (pre-surgery) and postoperative adjuvant therapy.
  Treatment Protocol
  Preoperative (4-6 cycles) and Postoperative (6-8 cycles):
  Each 14-day cycle includes:
  Oxaliplatin: 85 mg/m² via 180-minute intravenous infusion on Day 1.
  Leucovorin: 400 mg/m² via 120-minute intravenous infusion on Day 1.
  5-Fluorouracil: 2400 mg/m² via continuous intravenous infusion over 46 hours.
  Other Names: 5-Fluorouracil, Oxaliplatin
  Arms: mFOLFOX regimen neoadjuvant therapy group

SUMMARY:
This study is a prospective, open-label, two-arm, phase II clinical trial involving patients preoperatively diagnosed with YWHAB (Tyrosine 3-monooxygenase/tryptophan 5-monooxygenase activation protein beta)-high locally advanced rectal cancer. The trial evaluates a regimen combining mFOLFOX chemotherapy with citrus flavonoid tablets (Alvenor) for neoadjuvant therapy (pre-surgery) and postoperative adjuvant therapy.

Treatment Protocol

Preoperative (4-6 cycles) and Postoperative (6-8 cycles):

Each 14-day cycle includes:

Oxaliplatin: 85 mg/m² via 180-minute intravenous infusion on Day 1.

Leucovorin: 400 mg/m² via 120-minute intravenous infusion on Day 1.

5-Fluorouracil: 2400 mg/m² via continuous intravenous infusion over 46 hours.

Citrus flavonoid tablets (Alvenor) : 500 mg orally three times daily (Days 1-14), administered with or without the chemotherapy regimen (depending on group assignment).

Key Trial Design Features Dose Adjustments: Permitted during the trial based on patient tolerance.

Discontinuation Criteria:

Patients with disease progression during neoadjuvant therapy will cease study treatment and proceed to surgery or alternative therapies per local guidelines.

Surgery may be initiated early if patients cannot tolerate the planned 6 cycles of neoadjuvant therapy.

Patients receiving non-protocol anticancer therapies preoperatively will be withdrawn from the study.

Postoperative Management:

Post-treatment plans (e.g., continuation of mFOLFOX + Alvenor) are determined by the investigator.

Control Group Restriction: Patients in the control arm are not permitted to self-administer citrus flavonoid tablets (Alvenor) during the trial. Any requirement for this medication must be discussed with the treating physician, who will decide on alternative therapies or trial withdrawal.

DETAILED DESCRIPTION:
This study plans to conduct a prospective, open-label, two-arm, phase II clinical trial: For patients with locally advanced rectal cancer, YWHAB immunohistochemical staining will be performed on endoscopic biopsy specimens to screen out patients with high expression of YWHAB in locally advanced rectal cancer. These patients will be randomly assigned to the mFOLFOX treatment group or the mFOLFOX combined with Citrus Flavone Tablets (Alvenor) treatment group for neoadjuvant therapy. After completing 4-6 cycles of neoadjuvant chemotherapy, the patients will undergo preoperative assessment by the attending physician and surgical resection of the tumor by a professional colorectal surgery team. Postoperatively, they will receive 6-8 cycles of adjuvant chemotherapy. The efficacy (proportion of patients achieving tumor downstaging, three-year disease-free survival rate, overall survival time, and tumor regression grade TRG, etc.) and safety (drug-related adverse reactions, etc.) of the mFOLFOX combined with Citrus Flavone Tablets (Alvenor) neoadjuvant therapy for patients with high expression of YWHAB in locally advanced rectal cancer will be evaluated to assess the efficacy, safety, and feasibility of this treatment regimen. Based on the team's previous basic/translational research, animal experiments, and the clinical safety of Citrus Flavone Tablets (Alvenor), this study is expected to improve the efficacy of patients with high expression of YWHAB in locally advanced rectal cancer and benefit more patients.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed rectal adenocarcinoma: All other histological types are excluded. The patients have concurrent hemorrhoids documented by colonoscopy report or clinical physical examination.
* Clinical Pathological Stage: Tumor staged as T3-4 or N+, M0 (according to the AJCC （American Joint Committee on Cancer）TNM （Tumor-Node-Metastasis) Staging System, 9th Edition; see Appendix 1).
* Biomarker Status: Immunohistochemical staining of the tissue specimen demonstrates high expression of YWHAB in rectal cancer.
* Age: 18 to 75 years old, inclusive, at the time of signing the Informed Consent Form (ICF).
* Performance Status: Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (see Appendix 3).
* Prior Therapy: No prior systemic anti-tumor therapy for rectal cancer, including cytotoxic chemotherapy, immune checkpoint inhibitor therapy, molecular targeted therapy, endocrine therapy, etc.
* Adequate Organ Function: Based on laboratory values obtained during the screening period:White Blood Cell (WBC) count ≥ 3.0 × 10⁹/L, absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L, platelet count ≥ 75 × 10⁹/L, serum Total Bilirubin ≤ 1.5 × Upper Normal Limit (UNL), aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≤ 2.5 × UNL, serum Creatinine ≤ 1.5 × UNL.
* Contraception (Females of Childbearing Potential - FCBP): FCBP must have a negative serum pregnancy test within 3 days prior to initiation of study treatment. They must be willing to use a medically approved highly effective method of contraception (e.g., intrauterine device, oral contraceptives, condoms) during the study period and for 3 months after the last dose of study drug.
* Contraception (Males): Male subjects with partners of childbearing potential must use effective methods of contraception during the study period and for 3 months after the last dose of study drug.
* Consent and Compliance: The subject has voluntarily agreed to participate by signing the ICF and is willing and able to comply with scheduled visits, study treatment, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Distant Metastasis: Confirmed by systemic imaging (CT（Computed Tomography）, MR （Magnetic Resonance Imaging）, or PET-CT （Positron Emission Tomography - Computed Tomography）) encompassing at least the chest, abdomen, and pelvis.
* Pharmacogenetic Deficiency: Known complete DPD (dihydropyrimidine dehydrogenase) enzyme deficiency or homozygous UGT1A1*28 (7/7) genotype identified by whole-genome testing.
* Acute Surgical Complications: Presence of complete intestinal obstruction, active bleeding, or perforation requiring emergency surgery.
* Other Active Malignancies: History or concurrent presence of other active malignancies, except for malignancies treated with curative intent with no recurrence for >5 years, or adequately treated carcinoma in situ (e.g., cervical carcinoma in situ, non-melanoma skin cancer).
* Thromboembolic Events: History of thromboembolic events (e.g., cerebrovascular accident [including transient ischemic attack], pulmonary embolism, deep vein thrombosis) within 12 months prior to study enrollment.
* Significant Cardiac Disease: Occurrence of any of the following within 12 months prior to enrollment: myocardial infarction, severe/unstable angina, heart failure of NYHA （New York Heart Association Functional Classification）class 2 or higher, clinically significant supraventricular or ventricular arrhythmia requiring treatment, or symptomatic congestive heart failure.
* Recent Infection/Fever: Systemic antibiotic use for ≥7 days within 4 weeks prior to enrollment, or unexplained fever >38.5°C during screening or prior to the first dose (fever attributed to the tumor by the investigator is allowed).
* Major Surgery/Trauma: Undergone major surgery (e.g., laparotomy, thoracotomy, organ resection via laparoscopy) or experienced significant trauma within 2 months prior to enrollment. The surgical incision must be fully healed before study entry.
* HIV/AIDS: Known HIV (Human Immunodeficiency Virus) infection or AIDS (Acquired Immunodeficiency Syndrome)-related illness.
* Significant Pulmonary/Systemic Disease: Presence of interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (e.g., diabetes mellitus, hypertension, pulmonary fibrosis, acute pneumonitis).
* Untreated Active Hepatitis: Untreated active hepatitis B virus (defined as HBV-DNA ≥ 500 IU/mL) or hepatitis C virus (defined as HCV-RNA above the lower limit of quantification), or known co-infection with HBV and HCV.
* Drug Hypersensitivity: Known or suspected history of hypersensitivity to any of the drugs related to the study treatment.
* Investigator Discretion: Any other condition that, in the judgment of the investigator, would make the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Tumor downstaging rate (to ypTNM stage 0-I) | Perioperative，2 weeks after surgery
  The proportion of patients with locally advanced rectal cancer who, after receiving neoadjuvant chemotherapy with mFOLFOX or mFOLFOX plus Citrus flavonoid tablets (Alvenor), were downstaged to ypTNM stage 0-I based on postoperative surgical specimens.

SECONDARY OUTCOMES:
Three-year disease-free survival | through study completion, an average of 3 year
  Disease-free survival (DFS) was defined as the proportion of patients who, from the time of randomization until the end of year 3, did not experience any of the following events: disease progression; macroscopic or microscopic residual tumor after surgery; local recurrence; distant metastasis; or death from any cause, whichever occurred first.
Overall survival | through study completion, an average of 5 year
  Overall survival (OS) was defined as the time from randomization to death from any cause.
tumor regression grade (TRG) | Perioperative，2 weeks after surgery
  TRG 0 indicates no residual tumor cells; TRG 1 indicates single cells or small groups of cells; TRG 2 indicates residual cancer with a desmoplastic response; and TRG 3 indicates minimal evidence of tumor response.
Rate of Treatment-Related Adverse Events (Grade 3 or Higher) | through study completion, an average of 1 year
  Treatment-related adverse event rate (Grade ≥3): Refers to grade 3 or higher adverse drug reactions determined to be related to the investigational antineoplastic drug/treatment in clinical trials, excluding nonspecific infusion reactions.
Complete response (CR) rate | Perioperative，2 weeks after surgery
  The proportion of patients with complete response (CR) after surgery. Complete response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Partial response (PR) rate | Perioperative，2 weeks after surgery
  The proportion of patients with partial response (PR) after surgery. Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Stable disease (SD) rate | Perioperative，2 weeks after surgery
  The proportion of patients with stable disease (SD) after surgery. Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Progressive disease (PD) rate | Perioperative，2 weeks after surgery
  The proportion of patients with progressive disease (PD) after surgery. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (including the baseline if that is the smallest), with an absolute increase of at least 5 mm, or the appearance of one or more new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaosheng He, M.D./Ph.D, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT07176182/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT07176182/ICF_001.pdf